CLINICAL TRIAL: NCT06818825
Title: Point of ED Discharge Interactive Outreach: High ED Utilizers
Brief Title: Nudging High Emergency Department Utilizers to Consider Non-emergent Healthcare Resources
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-0686
Record Dates: First submitted 2025-01-29; First posted 2025-02-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Emergency Service, Hospital
MeSH Terms: conditions — Emergencies | interventions — Communication Devices for People with Disabilities; CD56 Antigen

STUDY DESIGN:
Masking Description: Patients will be aware of their own messages but will not be aware of other messages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Worker/Community Medical Assistant Outreach (Active Comparator): Patients will receive outreach from a community health worker or a community medical assistant, as is current standard practice, including guidance about ED-alternative resources to encourage care outside of the ED when appropriate.
  Interventions: Behavioral: Live outreach
- SMS Chatbot Messages (Experimental): Patients will be sent interactive SMS chatbot messages, including guidance about ED-alternative resources to encourage care outside of the ED when appropriate; patients will not receive outreach from a community health worker or community medical assistant.
  Interventions: Behavioral: Automated interactive messages

INTERVENTIONS:
Behavioral: Automated interactive messages — High ED utilizers will be sent SMS text messages guiding them through ED-alternative resources, with different guidance (including a follow-up phone call from a healthcare worker) depending on patient responses.
  Other Names: Text
  Arms: SMS Chatbot Messages
Behavioral: Live outreach — High ED utilizers will be called (and possibly visited) by a CHW/CMA guiding them through ED-alternative resources.
  Other Names: Call
  Arms: Community Health Worker/Community Medical Assistant Outreach

SUMMARY:
The goal of this campaign is to reduce unnecessary ED visits by providing patients who are high ED utilizers (with a visit of any acuity) with alternative resources to manage their health outside of the ED. In this campaign, patients will be randomized to receive one of two types of outreach following discharge aligned with the goal. Outreach may occur via (1) a phone call from a Geisinger Community Health Worker (CHW) or Community Medical Assistant (CMA); current standard practice or (2) an interactive chatbot message providing similar information and questions to those provided by the CHW/CMA. The study team will measure whether ED use differs across patients in different outreach conditions. The study team will also examine whether patients followed through on the message-specific calls to action in the messages differently across conditions.

ELIGIBILITY:
Inclusion Criteria:

* Geisinger Health Plan insurance or KACO membership
* Any PCP or no PCP
* Visit of any acuity
* 4 or more ED visits in the past 6 months

Exclusion Criteria:

* Institutionalized
* Cannot be contacted via the communication modality being used in the study (i.e., SMS), due to insufficient/missing contact information in the electronic health record or because the patient opted out
* Admitted to hospital
* Eloped from ED
* Left ED without being seen
* Deceased prior to messaging
* Qualifies for more intensive care management due to higher-level category of complexity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1553 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Return to ED (Y/N) | Within 120 calendar days following day of discharge
  Patient had a new Geisinger ED encounter after being discharged

OTHER OUTCOMES:
Successful Patient Contact (Y/N) - 3 days | Within 3 business days following day of discharge
  At least one successful contact between patient and a CMA, a CHW, or a representative at the monitoring center (Y/N)
Successful Patient Contact (Y/N) - 5 days | Within 5 business days following day of discharge
  At least one successful contact between patient and a CMA, a CHW, or a representative at the monitoring center (Y/N)
Time to Contact | Within 30 calendar days following day of discharge
  Time to successful patient contact by monitoring center, CMA, or CHW
Patient replied via SMS text (Y/N) to Artera chatbot | Within 7 calendar days following first Artera outreach
  Patient responded to the Artera chatbot at least once (Y/N)
ED Use (Y/N) | Within 30 calendar days following day of discharge
  Patient had a new Geisinger ED encounter after being discharged
ED Use After Outreach (Y/N) | Within 30 calendar days following day of outreach by Artera, CMA, or CHW
  Patient had a new Geisinger ED encounter after receiving outreach

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/25/NCT06818825/Prot_SAP_000.pdf